CLINICAL TRIAL: NCT02167984
Title: Esophageal Bolus Transit in GERD Newborns: a Multichannel Intraluminal Impedance Study
Brief Title: Esophageal Bolus Transit in Newborns With Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Francesco Cresi, MD, PhD, MD, University of Turin, Italy
Other Study IDs: swallow-01
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Gastroesophageal Reflux
Keywords: esophageal swallow; gastroesophageal reflux; esophageal impedance; newborn; preterm
MeSH Terms: conditions — Gastroesophageal Reflux; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- at term newborns: Infant with GE >=37w
- preterm newborns: Infant with GE <37w

SUMMARY:
Esophageal dysmotility due to immaturity could promote impaired bolus transit during esophageal swallow events,thus influencing gastroesophageal reflux (GER) clearance.

Aim of this study was to describe esophageal bolus transit characteristics during swallow and to evaluate the relationship between esophageal swallow (ES) and GER in newborns with gastroesophageal reflux disease symptoms using multichannel intraluminal impedance.

The simultaneous analysis of swallow and GER events in newborns undergone MII/pH monitoring could provide useful information to better understand the physiopathology of gastroesophageal reflux disease (GERD) and could help clinicians to identify newborns with prolonged esophageal clearance time, making the recommendations for further tests and the therapeutic approach more accurate

DETAILED DESCRIPTION:
The aim of this study was to evaluate esophageal swallow (ES) frequency and characteristics in term and preterm newborns with GERD symptoms using MII and to investigate the possible relationship between ES and GER events.

MATERIAL AND METHODS

The MII tracings from the beginning of the second feeding up to 3 hours after the end of the meal were visually analyzed by two independent investigators using Bioview Analysis software (Sandhill Scientific Inc., Highlands Ranch, Colorado, USA) to identify and characterize ES and GER events.

ES events An ES event was identified as a rapid increase in impedance which precedes a drop in impedance to 50% of baseline beginning in the proximal channel and preceding in an anterograde direction to the most distal channel, followed by the recovery of baseline values at each channel.13 The ES events detected by MII/pH were grouped into mealtime events (the first nine consecutive ES events with no artifacts after the beginning of the meal) and postprandial period events (all the ES events detected in the 3 hours following the end of the meal).

ES event frequency (ES events/hour) was measured, along with the following ES event characteristics:

bolus presence time (BPT): time between bolus entrance and exit recorded in the distal channel, measured in seconds; bolus head advancing time (BHAT): time between the bolus entrance recorded in the proximal channel and the bolus entrance recorded in the distal channel, measured in seconds; bolus head advancing time corrected (BHATc): BHAT corrected for esophageal length, expressed in seconds/cm. BHATc was calculated using the formula BHATc = BHAT / esophageal length where esophageal length is the distance between proximal and distal impedance channels, measured in cm.

GER events

A GER event was defined as a retrograde drop in impedance to 50% of baseline, beginning in the most distal channel and proceding to one or more proximal channels, of at least 5 seconds, followed by an impedance recovery of baseline values.GER event frequency was measured (GER events/hour), along with the following event characteristics:

bolus reflux extent (BRE):the proximal extent reached by the refluxate, shown by the number of channels sequentially involved in the impedance drop,measured in number of channels; bolus clearance time (BCT):time from onset, at the 50% drop in impedance signal from baseline, to the end of the event, at the 50% recovery point from nadir to baseline, recorded in the distal impedance channel, measured in second.

Statistical Analysis The distribution of all the continuous variables was assessed by the Shapiro-Wilk test. The differences in MII variables between different groups of infants were evaluated with the Mann-Whitney test; the Wilcoxon test was used to compare paired data. Group correlations were analyzedwith the Spearman correlation test. Statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentations included regurgitation/vomiting, apnea and desaturations, coughing, feed refusal, irritability, crying, back arching, failure to thrive.

Exclusion Criteria:

* Presence of congenital abnormalities, perinatal asphyxiation or neurological pathologies Taking drug known to influence esophageal motor function. Anti-reflux treatment was ceased 1 week before MII/pH.

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborns consecutively admitted to the Torino University NICU who underwent 24-hour MII/pH for suspected GERD
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
BPT, BHAT, BHATc | calculated throughout 24 hours
  bolus presence time (BPT): time between bolus entrance and exit recorded in the distal channel, measured in seconds; bolus head advancing time (BHAT): time between the bolus entrance recorded in the proximal channel and the bolus entrance recorded in the distal channel, measured in seconds; bolus head advancing time corrected (BHATc): BHAT corrected for esophageal length, expressed in seconds/cm. BHATc was calculated using the formula BHATc = BHAT / esophageal length

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cresi, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Ospedale OIRM - S.Anna di Torino, Torino, (TO), Italy

IPD SHARING:
Plan to Share IPD: No